CLINICAL TRIAL: NCT04599205
Title: Evaluation of Fractional CO2 Laser and Tranexamic Acid in Treatment of Melasma:Clinical,Histopathological and Immunohistochemical Study
Brief Title: Evaluation of Laser and Tranexamic Acid in Treatment of Melasma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Hasan, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOFCLATAITOMCHAIS
Record Dates: First submitted 2020-09-09; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid; Lasers; Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Microneedling group A (Experimental): Patients will be subjected to the following:
  Combined laser (power=3.6 mJ) and topical tranexamic acid (TXA) (one finger unit) gel on the right half of the face.
  Combined microneedling (by dermapen) and topical TXA gel only on the left half. Self application of topical TXA gel (2 finger units) on both sides on daily base.
  Interventions: Drug: Tranexamic acid
- Laser group B (Experimental): Patients will be subjected to the following:
  Combined laser(power=3.6 mJ) and topical TXA gel (one finger unit) on the right half.
  Laser (power=3.6 mJ) only on the left one.
  Interventions: Drug: Tranexamic acid
- Gel group C (Experimental): patients will be subjected to: Daily application of topical TXA gel (2 finger units) on both face sides.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — fractional co2 laser, microneedling and topical tranexamic acid gel
  Other Names: laser; microneedling

SUMMARY:
Melasma Is an acquired, chronic, recurrent, symmetrical hypermelanosis, which is characterized by brown patches of variable darkness on sun exposed areas of the body. It is more common in women. It is common psychologically and emotionally distressing cosmetic problem in affected patients .

DETAILED DESCRIPTION:
Many studies examined multiple treatment options for melasma , but none of them is completely satisfactory with recurrence in most cases.

Tranexamic acid is is a relatively new drug for melasma . It is currently used via a spectrum of delivery routes including oral, topical, intradermal, and microneedling .

Laser-assisted drug delivery (LADD) is a technique that facilitates the delivery of topical medications .

On reviewing the previous literatures, few studies have focused on therapeutic effects of combined laser and TXA (topical and intradermal) in melasma, with variations in parameters of laser, in dose, concentration, form and routes of TXA application; and in follow up duration. These studies revealed variable unproven results, and since melasma is a challenging disease, additional studies are needed to determine the optimal laser parameters and the best absorbable topical TXA formula, ensuring the best efficacy and less complications.

To the best of our knowledge, this is the first study that will use topical TXA gel as an additive effect between sessions, and to confirm the effect of laser and TXA by histopathology and immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* - Gender: Only female patients.
* Age: 18-50 years old.
* Type of melasma: Bilateral symmetrical facial melasma of all types.
* Fitzpatrick skin phototypes: Types III, IV and V.

Exclusion Criteria:

* - Pregnancy and lactation.
* Patients taking oral contraceptive pills, hormonal replacement therapy or isotretinoin at the time of the study or during the past 6 months. Concomitant use of anticoagulants, bleeding disorders.
* Scarring and keloid tendency, active skin infections, active HSV, and those with facial cancer.
* History of photosensitivity or photosensitizing medications such as sulfonamides and tetracycline.
* Previous history of post inflammatory hyperpigmentation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
safety and effectiveness of fractional CO2 laser, microneedling and topical tranexamic acid gel | 2 years
  the therapeutic effect of combined fractional co2 laser and topical tranexamic acid versus either fractional co2 laser alone, topical TXA alone or combined microneedling and TXA in treatment of melasma.this will be assessed by melasma area and severity index (MASI).

SECONDARY OUTCOMES:
accurate outcome of each treatment modality | 2 years
  every modality's effect will be measured by the histopathological changes by use of fontana asson stain.

CONTACTS AND LOCATIONS:
Overall Officials: EMAN R MOHAMED, MD, Study Director — assuit university hospital

IPD SHARING:
Plan to Share IPD: No